CLINICAL TRIAL: NCT01580722
Title: Study of Surgical Methods for Anterior Cruciate Ligament Tearing
Brief Title: Comparison of Early Versus Delay Reconstruction in Anterior Cruciate Ligament Tearing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamidreza Shemshaki, principle, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASD-1213-100
Record Dates: First submitted 2012-04-18; First posted 2012-04-19 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Anterior Cruciate Ligament Tear
Keywords: Anterior Cruciate Ligament,Early,Delay,Reconstruction
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- early (Other): patients underwent < 8 weeks reconstruction after injury
  Interventions: Procedure: early reconstruction
- delay (Other): patients underwent > 8 weeks reconstruction after injury
  Interventions: Procedure: delay reconstruction

INTERVENTIONS:
Procedure: early reconstruction — patients underwent < 8 weeks reconstruction after injury
  Arms: early
Procedure: delay reconstruction — patients underwent > 8 weeks reconstruction after injury
  Arms: delay

SUMMARY:
The purpose of this study is to determine which surgical method is better for anterior cruciate ligament teas in outcomes.

DETAILED DESCRIPTION:
The anterior cruciate ligament (ACL) is one of the most commonly injured ligaments of the knee. This study was conducted to determine whether the outcome of treatment is superior in early surgical reconstruction compared with optional delay reconstruction.

ELIGIBILITY:
Inclusion Criteria:

a. patients with confirmed anterior cruciate ligament tearing

Exclusion Criteria:

One of the following associated injuries to the index knee as visualized on MRI and/or arthroscopy:

1. An unstable longitudinal meniscus tear that requires repair and where the following postoperative treatment (i.e. bracing and limited ROM) interferes with the rehabilitation protocol
2. Bi-compartmental extensive meniscus resections
3. A cartilage injury representing a full thickness loss down to bone
4. A total rupture of MCL/LCL as visualized on MRI

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2012-03; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
quality of life | at 6 months post-operatively
  SF-36 questionnaire consists of 36 questions (two main components: physical and mental), each of which was assigned a score ranging from 0 to 100.

SECONDARY OUTCOMES:
Tegner activity score | at 6 months post-operatively
  The Tegner Activity Scale depicts the level of sporting activity and allows us to compare and document the preinjury activity level with the present activity level. This numeric score ranging from 1 to 10 where 1 is the least strenuous activity for the knee and 10 is the hardest.
Knee injury and Osteoarthritis Outcome Score | at 6 months post-operatively
  The Knee injury and Osteoarthritis Outcome Score is the extended form of The Western Ontario and McMaster Universities Arthritis Index (WOMAC) with 42 - items in 5 subscales consisting : pain ( 9 items ) , other symptoms ( 7 items ) , activities of daily living ( 17 items ) , sports and recreational function ( sport / rec ) ( 5 items ) , and knee - related quality of life ( QOL ) ( 4 items ) .

CONTACTS AND LOCATIONS:
Overall Officials: hamidreza shemshaki, MD, Study Chair — MD,research comittee
Locations (1):
- Al-zahra university hospital, Isfahan, Isfahan, Iran